CLINICAL TRIAL: NCT01130454
Title: A Double-blind Placebo-controlled Study of the Application of the SCIO Universal Electrophysiological Biofeedback System for Statistical Evaluation of the SCIO's Ability to Increase Body Wellness After One 45-minute Session
Brief Title: A Study for Evaluating the SCIO Biofeedback Device's Ability to Increase Body Wellness After One 45-minute Session
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maitreya Kft. (Industry)
Responsible Party: Richard Lloyd Regulatory Manager, Maitreya Kft
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-103-01
Record Dates: First submitted 2010-05-10; First posted 2010-05-26 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Stress
Keywords: Unfavorable effect of environmental factors, stressors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SCIO Test Group (Active Comparator)
  Interventions: Device: Universal Electrophysiological Biofeedback Treatment
- SCIO Placebo Group (Placebo Comparator)
  Interventions: Device: Universal Electrophysiological Biofeedback Treatment

INTERVENTIONS:
Device: Universal Electrophysiological Biofeedback Treatment — one 45 minute biofeedback treatment
  Other Names: SCIO biofeedback treatment
  Arms: SCIO Test Group
Device: Universal Electrophysiological Biofeedback Treatment — one 45 minute placebo treatment
  Other Names: placebo treatment
  Arms: SCIO Placebo Group

SUMMARY:
The objective of the study is to determine if one 45-minute treatment with the SCIO (Scientific Consciousness Interface Operations System) biofeedback device would show a change, and hopefully an improvement, on a person's Body Wellness indicators (Quality of Life Questionnaire, Energy Index Factor, Strength, Oxidation, Flexibility, Memory, pH, and VARHOPE scores (V=voltage, A=amperage, R=resistance, H=hydration, O=oxygenation, P=proton pressure and E=electron pressure), electrical measures within the device. For subjects in the control group, it is expected that there will likely be an improvement of approximately 5% in measured variables. That is, subjects in the control group will likely report some of the positive changes listed above for test group subjects. However, on average, any positive change in post-treatment measures for control subjects is expected to occur to a significantly lesser degree than for subjects in the test group.

DETAILED DESCRIPTION:
The objective of the Study is to determine if one 45-minute treatment with the SCIO (Scientific Consciousness Interface Operations System) biofeedback device would show a change, and hopefully an improvement, on a person's Body Wellness indicators as defined by the following introductions to each hypothesis. There are three (3) hypotheses that are the objective of this study and they are defined below as Hypothesis#1, Hypothesis#2 and Hypothesis#3.

Introduction#1: The body is an electrical process requiring volts and amps which conduct through resistance circuits to operate. All muscles are turned on by electrical impulse. Muscles themselves are magnetic using volts and amps for their operation. The brain is a massive collection of cells that have electrical activity that can be measured via the EEG (electroencephalography). The heart itself is the largest electro-magnetic engine and uses electrical impulses to influence the muscles of the heart to circulate blood. Most EEG (electroencephalography), ECG (electrocardiography) and EMG (electromyography) measures are only concerned with oscillatory properties and not so concerned with the volume or basic amperage of the circuit. The collective baseline of the circuit of EEG (electroencephalography), ECG (electrocardiography), EMG (electromyography) and GSR (galvanic skin response) measurements can give us a rating of the global body voltage, body amperage and skin resistance (V=voltage, A=amperage, and R=resistance respectively). There are norms of the V (voltage), A (amperage) and R (resistance) and certain people, due to stress or other factors, can have low V (voltage), A (amperage) and/or R (resistance).

Hypothesis#1: Our hypothesis is that by measuring and calculating the Voltage, Amperage and Resistance, and then administering one 45-minute treatment with the SCIO (Scientific Consciousness Interface Operations System) for stress reduction and electro-stimulation biofeedback, the Voltage, Amperage and Resistance can be rectified. Our scale is from 0-110 for the V, A and R measurements, so an improvement in these Body Wellness indicators is going towards the higher end of the scale.

Introduction#2: The collective inductance and capacitance changes in the body are a reflection of redox potential and can reflect hydration (H) and oxygenation (O) indexes.

Hypothesis#2: It is also the hypothesis of the study that these hydration (H) and oxygenation (O) indexes can be affected by one 45-minute treatment of stress reduction and the electro-stimulation biofeedback by the SCIO. Our scale is from 0-110 for the H and O measurements, so an improvement in these Body Wellness indicators is going towards the higher end of the scale.

Introduction#3: Irregularities in EEG, EMG, ECG and GSR can be corrected through guided electro-stimulation. The V and A are also greatly affected by the charge stability of the free protons and electrons, (negative charges and positive charges in the body), which collectively make up the proton pressure (P) and electron pressure (E). The acidity-alkalinity balance is an electrical measure of the amount of positive versus negative charged particles. This can be measured by the carbon based electrodes of the SCIO through electro-stimulation biofeedback.

Hypothesis#3: It is our hypothesis, that the proton pressure (P) and electron pressure (E) scores can be improved with one 45-minute treatment with the SCIO. The scale of normal P is 75 and the scale for normal E is 65 and the scores show an improvement in these Body Wellness indicators is if they change towards this number.

Together, these items of voltage (V), amperage (A), resistance (R), hydration (H), oxygenation (O), proton pressure (P) and electron pressure (E) form the term VARHOPE. These VARHOPE scores are essential for all body functioning, therefore our overall hypothesis is that within one 45 minute session, a measurable improvement in Body Wellness indicators can be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Individuals in this study will be humans who present with awareness of levels of perceived stress as well as injuries/pain as indicated by a response on the pre-test Wellness Questionnaire.
* Between 18 and 65 years of age.
* Male or female.

Exclusion Criteria:

* Extremely sick patients on more than 5 prescribed drugs
* Patients who are crippled, handicapped, or unable to move freely based on a licensed healthcare practitioner's statement
* Extremely healthy sports people or athletes with no symptoms or problems whatsoever
* Any known heart condition(s), such as cardiac arrhythmias, congestive heart failure disease, myocardial infarction
* Serious head trauma
* Pregnant, breast feeding, or planning pregnancy prior to the end of study participation
* Currently using a pacemaker
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in past two years
* Prior cardiac surgeries such as cardiac bypass, heart transplant surgery, pacemakers
* Seizure disorder or family history of seizure disorder
* Infection or wound or any other external trauma in the areas to which the electrode bands of the SCIO device are to be attached
* Developmental disability or cognitive impairment that would make it difficult for the subject to partake in the clinical study, including adequate comprehension of the informed consent form and ability to record the necessary measurements
* Involvement in litigation and/or a worker's compensation claim and/or receiving disability benefits because of a stress-related or involved condition
* Participation in a clinical study or other type of research in the past 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
VARHOPE Score | average 3 months
  VARHOPE is an acronym coined by the manufacturer in which V = Voltage, A = Amperage, R = Resistance, H = Hydration, O = Oxygenation, P = Protons and E = electrons.
  The VARHO readings are set on a scale from 0-110. Changes in the readings are shown on the scale where an increase in number shows in improvement.
  The PE readings are set on a scale where the closer the P reading to 75 the more the client's state of wellness has stabilized, and the closer the E reading to 65 the more the client's state of wellness has stabilized.

SECONDARY OUTCOMES:
Energy Index Factor | average 3 months
  Measurements taken: blood pressure and pulse left arm sitting.
  The Energy Index Factor formula used:
  Take the systolic left arm sitting + the diastolic left arm sitting x pulse = energy index factor.
  * Below 9,000 indicates parasympathetic control.
  * 14,000 indicate balance.
  * 18,000+ indicate sympathetic neural control.
Strength Test | average 3 months
  Patient holds the Dynamo-meter in one hand. They give one big squeeze with one hand on the Dynamo-meter and the investigator documents how many kilograms of strength the patient was able to exert. Done for both left and right hand.
Anaerobic Oxygenation Test | average 3 months
  Patient starts in a seated position, relaxed and at a normal breath rate for 1 minute. The patient takes a deep breath at the same time that the investigator starts a stop-watch counting minutes, seconds and tenths-of-a-second. Patient stands up at a normal speed and sits down again at a normal speed while still holding breath as long as possible. As soon as patient stops holding breath and takes a new breath then investigator stops the stop-watch. Investigator must document the length of time that the patient held breath during Anaerobic Oxygenation Test.
Low Back Flexibility | average 3 months
  Patient sits on the floor with legs stretched out in front, heels approximately 8 inches apart. The patient extends both hands, outstretched fingers towards their heels keeping legs straight. Patients are asked to do maximum stretch and touch the floor as far as they can, even going past the heels, if they can. The distance in inches from where their fingers touched the floor to the heels, with Zero at the heels, positive if they can extend past the heels, minus if they are before the heels. Normal scores are anywhere from -3 to 0, scores below -3 indicate low back difficulty.
Side to Side Flexibility | average 3 months
  Patient stands on their knees without bending forward or backward at the waist, they lean to the left side and try to touch their left palm to the floor. Touch their knuckles to the floor or try to touch their fingers to the floor and we measure the extent of their flexibility. Normal readings are touching fingers or knuckles to floor. An advanced patient will be able to touch their palm. If they cannot touch their fingers it indicates a lack of flexibility. A protractor is used to determine the angle of flexibility.
Neck Flexibility | average 3 months
  Patient tries to touch their ear to their shoulder without raising their shoulder to their ear. A protractor is used to determine the angle of flexibility.
Memory Test | average 3 months
  A series of random digits is chosen. The suggested test method is to choose the first set of random numbers. If the patient remembers these numbers in the proper sequence (either forward or backward depending on the memory test), then the investigator adds 2 to the existing digit and adds one more digit to the end to increase the sequence by one digit. This method should be continued until the end. The investigator should always write down the digit to ensure that they can reference the actual list when the patient repeats the digits.
pH Test | average 3 months
  An Over-The-Counter pH (acidity-alkalinity) Test Kit should be purchased and used for pre-test and post-test measurements. The pre-test reading should be taken within three (3) hours before the Treatment begins. The post-test may not be taken more than three (3) hours after the Treatment is completed.
Quality of Life Questionnaire | average 3 months
  The investigator asks the patient the following questions. The Investigator explains that the rating is on a scale of 1-10, where 10 is more negative and 1 is more positive.
  1. Rate your stress level.
  2. Rate how you feel in general.
  3. Do you have pain? Circle one: Yes/No. If yes, rate your pain.
  4. Do you have emotional trauma? Circle one: Yes/No. If yes, rate your trauma.
  5. Do you have an injury that causes discomfort? Circle one: Yes/No. If yes, rate your injury.
  6. Rate any symptoms you have that are of concern.

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Mutschler, MD, Principal Investigator
Locations (4):
- Annex of Quantum Northwest Presents, Seattle, Washington, United States
- Annex of Hexagram SARL, Paris, France
- CFI Centrum für Integrative Medizin, Speyer, Germany
- Centrul de Biorezonanţă Dr. Băcean, Timișoara, Timiș County, Romania